CLINICAL TRIAL: NCT03752918
Title: The Effects of MDMA on Prefrontal and Amygdala Activation in Posttraumatic Stress Disorder
Brief Title: The Effects of MDMA on Prefrontal and Amygdala Activation in PTSD.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding ended.
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Benjamin Kelmendi, MD, Associate Research Scientist, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000020348
Record Dates: First submitted 2018-11-16; First posted 2018-11-26 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: MDMA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Niacin

STUDY DESIGN:
Intervention Model Description: This study will be a double-blind, placebo-controlled, within-subjects, crossover-dose neuroimaging study in which participants will initially receive either a single dose of MDMA 1.5mg/kg or a placebo (niacin 250mg), with a crossover dose to follow. Doses will be separated by 2 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MDMA (Experimental): MDMA (1.5mg/kg)
  Interventions: Drug: MDMA
- Niacin (Placebo Comparator): Niacin (250mg)
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: MDMA — A single dose of 1.5mg/kg will be administered once orally.
  Other Names: 3,4-Methylenedioxymethamphetamine
  Arms: MDMA
Drug: Niacin — A single dose of 250mg will be administered once orally.
  Other Names: Nicotinic acid
  Arms: Niacin

SUMMARY:
This study aims to investigate the effects of MDMA on prefrontal and amygdala activation, and to explore the relationship between these MDMA-induced neural changes and the acute behavioral effects of the drug in patients with PTSD.

DETAILED DESCRIPTION:
The investigators intend to utilize state-of-the-art validated Human Connectome Project (HCP) style approaches to determine the effects of MDMA on prefrontal and amygdala activation, and to explore the relationship between these MDMA-induced neural changes and the acute behavioral effects of the drug in patients with PTSD. In addition, the investigators will collect preliminary data on the MDMA effects on large-scale intrinsic functional connectivity using novel graph-based network analyses.

Specifically, the investigators will measure medial prefrontal cortex (mPFC) and amygdala activation in response to negative stimuli in patients with PTSD. The investigators hypothesize that MDMA will increase mPFC, but decrease amygdala, activation in response to negative stimuli.

The investigators will also explore the relationship between the MDMA-induced mPFC and amygdala activation, and performance on Ekman's Emotional Facial Expression task. This task is modulated by the mPFC and amygdala and as well as trauma severity in participants with PTSD. And finally, to explore the effects of MDMA on resting-state functional connectivity (rs-fcMRI) the investigators will use Coupled Intrinsic Connectivity Distribution (Coupled-ICD); an innovative, graph-based, fully data-driven approach that is particularly sensitive to paired rs-fcMRI data (e.g. pre/post-treatment).

Adult participants with PTSD will be recruited for a double-blind, placebo-controlled, within-subjects, crossover-dose neuroimaging study in which they will initially receive either a single dose of MDMA 1.5mg/kg or a placebo (niacin 250mg), with a crossover dose to follow. Doses will be separated by 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 21-55 years. Females will be included if they are not pregnant and agreed to utilize a medically (non-hormonal)* accepted birth control method (to include implant birth control, condom, diaphragm with spermicide, intrauterine device, tubal ligation, abstinence, or partner with vasectomy) or if post-menopausal for at least 1 year, or surgically sterile.
* Able to provide written informed consent according to Yale HIC guidelines.
* Able to read and write English as a primary language.
* Diagnosis of PTSD, as determined by the Clinician Administered PTSD Scale (CAPS-5).
* Must have a score of 23 or higher on the Clinician-Administered PTSD Scale (CAPS-5) at screening.
* No more than mild TBI according to a modified version of the Brief TBI Screen.
* Must not have a medical/neurological problem or use medication that would render MDMA unsafe by history or medical evaluation.
* No prior exposure to MDMA.
* Are willing to remain overnight at the study site after each experimental session.
* Are willing to be driven home the day after the experimental sessions.
* Not currently taking any of the listed medications at the time of the study.
* Are willing to sign a medical release for the investigators to communicate directly with their therapist and doctors.
* Are willing to abstain from alcohol, street drugs, and tobacco products while in the study.

Exclusion Criteria:

* Patients with a diagnostic history of bipolar disorder, schizophrenia or schizoaffective disorder or currently exhibiting psychotic features as determined by the MINI 7.0 for the DSM-5.
* Serious suicide or homicide risk, as assessed by evaluating clinician.
* Substance abuse or dependence during the 6 months prior to screening; or a positive pre-study (screening) urine drug screen.
* Any significant history of serious medical or neurological illness.
* Any signs of major medical or neurological illness on examination or as a result of ECG screening or laboratory tests (e.g. positive urine tox, positive HIV/AIDS tests ).
* Abnormality on physical examination. A participant with a clinical abnormality may be included only if the study physician considers the abnormality will not introduce additional risk factors and will not interfere with the study procedure.
* Pregnant or lactating women or a positive urine pregnancy test for women of child-bearing potential at screening or prior to any imaging day.
* Any history indicating learning disability, mental retardation, or attention deficit disorder.
* Family history of cardiovascular diseases. History of hypertension with baseline blood pressure above 140 mmHg (systolic) and over 90 mmHg (diastolic). Any history of syncope and/or baseline blood pressure below 100mmHg (systolic).
* History of claustrophobia.
* BMI > 30 kg/m2 or >250 pounds.
* Anxiolytic, neuroleptic and SRI medications (off SRIs for 4 weeks, fluoxetine 5 weeks).
* Females taking hormonal contraceptives will not be able to participate in the study *(Hormonal contraceptives are exclusionary because MDMA increases production of oxytocin which is heavily modulated by other hormones (e.g. estrogen). Therefore, women need to be naturally cycling/ovulating and not taking any hormonal medications to participate in this study).
* Any metal or electromagnetic implants, including: (Cardiac pacemaker, artificial heart valve, defibrillator, aneurysm clip, cochlear implants, shrapnel, neurostimulators, history of metal fragments in eyes or skin, significant hearing loss or other severe sensory impairment, a history of seizures or current use of anticonvulsants.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Changes in activation of mPFC, amygdala, and nucleus accumbens upon presentation of emotional faces. | Initial Drug Dose, 2 weeks post drug dose (second drug dose).
  This will be assessed using mixed effects regression models, with group, time, and group X time effects modeled to examine the effect of MDMA on region of interests (ROI) activation. We will also assess the functional connectivity of between these ROIs.

SECONDARY OUTCOMES:
Changes in PTSD symptoms, which will be measured by The Clinician-Administered PTSD Scale 5 (CAPS-5). | Baseline, Initial Drug Dose and Second Drug Dose, 24 hours and 1 week after initial and second drug dose.
  Assesses PTSD symptoms. It is a structured interview that consists of 30 items. Items are rated using a 0 to 4 severity scale. In addition to assessing the 20 DSM-5 PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization. Higher scores indicate more severe PTSD symptoms.
Changes in depression symptoms, which will be measured by The Beck Depression Inventory II (BDI-II). | Baseline, Initial Drug Does and Second Drug Dose, 24 hours after initial and second drug dose, 3 and 5 days after initial and second drug dose (by phone), 1 week after initial and second drug dose, 15, 17, 19, and 21 days after second drug dose (phone).
  Assesses depression symptoms. Consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression.
Changes in sleep patterns, which will be measured by The Pittsburgh Sleep Quality Index (PSQI). | Baseline, 24 hours after first and second drug dose, 1 week after initial and second drug dose.
  Assesses the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. Items are rated using a 0 to 3 scale. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Changes in PTSD symptoms, which will be measured by The Posttraumatic Stress Disorder Checklist for the DSM-5 (PCL-5). | Baseline, 24 hours after initial and second drug dose, 3 and 5 days after initial and second drug dose (phone), 1 week after initial and second drug dose, 15, 17, 19, and 21 days after second drug dose (phone).
  Assesses PTSD symptoms. It is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Items are rated using a 0 to 4 scale. Total scores range from 0 to 80, with higher scores indicating more severe PTSD symptoms.
Changes in personality traits, which will be measured by The NEO Personality Inventory - Revised (NEO PI-R). | Baseline, 1 week after initial and second drug dose.
  Assesses changes in personality traits. It is a personality inventory that examines a person's Big Five personality traits. It consist of 240 items that assess 30 specific traits, which in turn define the five factors: Neuroticism (N), Extraversion (E), Openness to Experience (O), Agreeableness (A), and Conscientiousness (C). Items are rated on a five-point Likert scale, from strongly disagree to strongly agree.
Changes in mental states, which will be measured The 5-Dimensional Altered States of Consciousness Scale (5D-ASC). | Initial and second drug dose.
  Assesses different mental states induced by the interventions. Consists of 94 items which are rated by placing marks on a horizontal visual analogue scale (100 millimeters in length). The scale ranges from no, not more than usual (on the left) to yes, very much more than usual (on the right). The items are scored by measuring the millimeters from the low end of the scale to the participant's mark (from 0 to 100).
Changes in growth following a traumatic event, which will be measured by The Post traumatic Growth Inventory (PTGI). | Baseline, 24 hours after initial and second drug dose, 1 week after initial and second drug dose.
  Assesses positive outcomes reported by persons who have experienced traumatic events. It is a 21-item scale that includes factors of New Possibilities, Relating to Others, Personal Strength, Spiritual Change, and Appreciation of Life. Participants are asked to rate the degree to which this change occurred in their life as a result of the crisis/disaster. Each item is rated from 0 (I did not experience this change as a result of my crisis) to 5 (I experienced this change to a very great degree as a result of my crisis). Total score is calculated by summing all items. Individual factors are scored by adding responses to items on each factor. Higher scores indicate greater growth.
Changes in well-being, which will be measured by The Well-Being Inventory (WBI). | Baseline, 1 week after initial and second drug dose.
  Assesses well-being across life domains and such as work, finances, health, and social relationships. Participants are first asked questions about their level of functioning in each domain. Items are rated from 1 (never) to 5 (most or all of the time). Then they are asked questions about their satisfaction in each domain. Items are rated from 1 (very dissatisfied) to 5 (very satisfied). Higher total scores indicate greater well-being.
Changes in psychological inflexibility/experiential avoidance, which will be measured by The Acceptance and Action Questionnaire II (AAQ-II). | Baseline, 1 Week after initial and second drug dose.
  Assesses psychological inflexibility/experiential avoidance. Participants are asked to rate how true each statement is for them. Items are rated from 1 (never true) to 7 (always true). Higher scores equal greater levels of psychological inflexibility.
Changes in emotional regulation, which will be measured by The Emotion Regulation Questionnaire (ERQ). | Baseline, 1 week after initial and second drug dose.
  Assesses emotional regulation. A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Participants answer each item on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The higher the scores the greater the use of the emotion regulation strategy.
Changes in cognitive and emotional empathy, which will be measured by the Multifaceted Empathy Test (MET). | Baseline, Initial and Second Drug Dose, 24 hours after initial and second drug dose, 1 week after initial and second drug dose.
  Measures cognitive and emotional empathy simultaneously and independently using a series of photorealistic stimuli computer based tasks.
Changes in the quality of specific relationships in terms of supportive and conflictual dynamics will be assessed with the Quality of Relationships Inventory (QRI) | Baseline, Initial and Second Drug Dose, 1 week after initial and second drug dose.
  The 25 question task assesses the contemporary quality of specific relationships (between the patient and a specific individual, such as a family member) at a particular point in time in terms of conflict, support, and depth. It uses a Likert-type 4 point scale going from "1" indicating the item does not apply at all, while "4" indicates the item applies quite a lot.
Cognitive schemas about oneself and others, will be assessed by the Trauma and Attachment Beliefs Scale (TABS) | Baseline
  The 84 item self-report scale, which measures responses on a 1-6 scale (1 = "Disagree Strongly, 6 = Agree Strongly) the degree to which respondents believe the statements correspond with their own beliefs. The measures of these beliefs relate to self-safety, other-safety, self-trust, other-trust, self-esteem, other-esteem, self-intimacy, other-intimacy, self-control, and other control.
Brain injury will be assessed for with the CogState Neuropsychological Test | Baseline, 1 week after initial and second drug dose.
  Brain injuries associated with traumatic events, such as concussions, will be screened for in the CogState Neuropsychological Test, a standard computerized test used to assess neuropsychological deficits associated with brain injury.
Moral injury, or the sense of distress due to contradiction of deeply-held beliefs due to a traumatic event, will be measured by the Moral Injury Events Scale (MIES) | Baseline, Initial and Second Drug Dose, 24 hours after initial and second drug dose, 1 week after initial and second drug dose.
  This 9 item self-report scale measures the moral injury, or distress due to the contradiction to a deeply-held belief about the world that often accompanies a traumatic incident. The injury is assessed in terms of "perceived transgression" and "perceived betrayal." Items are assessed with a Likert-type Scale (1 to 6, 1 = "strongly disagree," 6 = "strongly agree," with no neutral option). Higher scores indicate greater severity of associated event.
Changes in concept and sense of existential meaning will be measured with the Purpose and Meaning scale (PIL) | Baseline, 1 week after second drug dose.
  Measures evaluation of the sense of existential purpose and enthusiasm for life in a three part self-report survey. Part A is a 20 point scale test which uses a 1-7 scale in which low number answers correspond attitudes such as boredom and directionless-ness. Parts B and C are not empirically useful, but ask for participants to completes sentences and compose a paragraph respectively. Higher scores indicate a greater existential sense of purpose, with scores above 113 indicate a high degree of purpose, scores below 92 suggesting a lack of purpose, and scores between 92 and 112 indicate moderate levels of purpose.
Changes in depression symptoms, which will be measured Montgomery-Asberg Depression Rating Scale (MADRS). | Baseline, Initial and Second Drug Dose, 24 hours after initial and second drug dose, 1 week after initial and second administration.
  Assesses depression symptoms. Consists of 10 items and uses a 0 to 6 severity scale. Total scores range from 0 to 60, with higher scores indicating more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kelmendi, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haagen JF, Smid GE, Knipscheer JW, Kleber RJ. The efficacy of recommended treatments for veterans with PTSD: A metaregression analysis. Clin Psychol Rev. 2015 Aug;40:184-94. doi: 10.1016/j.cpr.2015.06.008. Epub 2015 Jun 27. PMID 26164548
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Pitman RK, Rasmusson AM, Koenen KC, Shin LM, Orr SP, Gilbertson MW, Milad MR, Liberzon I. Biological studies of post-traumatic stress disorder. Nat Rev Neurosci. 2012 Nov;13(11):769-87. doi: 10.1038/nrn3339. Epub 2012 Oct 10. PMID 23047775
- [Background] Abad S, Camarasa J, Pubill D, Camins A, Escubedo E. Adaptive Plasticity in the Hippocampus of Young Mice Intermittently Exposed to MDMA Could Be the Origin of Memory Deficits. Mol Neurobiol. 2016 Dec;53(10):7271-7283. doi: 10.1007/s12035-015-9618-z. Epub 2015 Dec 21. PMID 26687233
- [Background] Mithoefer MC, Wagner MT, Mithoefer AT, Jerome L, Doblin R. The safety and efficacy of +/-3,4-methylenedioxymethamphetamine-assisted psychotherapy in subjects with chronic, treatment-resistant posttraumatic stress disorder: the first randomized controlled pilot study. J Psychopharmacol. 2011 Apr;25(4):439-52. doi: 10.1177/0269881110378371. Epub 2010 Jul 19. PMID 20643699
- [Background] Mithoefer MC, Wagner MT, Mithoefer AT, Jerome L, Martin SF, Yazar-Klosinski B, Michel Y, Brewerton TD, Doblin R. Durability of improvement in post-traumatic stress disorder symptoms and absence of harmful effects or drug dependency after 3,4-methylenedioxymethamphetamine-assisted psychotherapy: a prospective long-term follow-up study. J Psychopharmacol. 2013 Jan;27(1):28-39. doi: 10.1177/0269881112456611. Epub 2012 Nov 20. PMID 23172889
- [Background] Shin LM, Rauch SL, Pitman RK. Amygdala, medial prefrontal cortex, and hippocampal function in PTSD. Ann N Y Acad Sci. 2006 Jul;1071:67-79. doi: 10.1196/annals.1364.007. PMID 16891563
- [Background] Shin LM, Liberzon I. The neurocircuitry of fear, stress, and anxiety disorders. Neuropsychopharmacology. 2010 Jan;35(1):169-91. doi: 10.1038/npp.2009.83. PMID 19625997
- [Background] Lanius RA, Bluhm R, Lanius U, Pain C. A review of neuroimaging studies in PTSD: heterogeneity of response to symptom provocation. J Psychiatr Res. 2006 Dec;40(8):709-29. doi: 10.1016/j.jpsychires.2005.07.007. Epub 2005 Oct 7. PMID 16214172
- [Background] Etkin A, Wager TD. Functional neuroimaging of anxiety: a meta-analysis of emotional processing in PTSD, social anxiety disorder, and specific phobia. Am J Psychiatry. 2007 Oct;164(10):1476-88. doi: 10.1176/appi.ajp.2007.07030504. PMID 17898336
- [Background] Carhart-Harris RL, Wall MB, Erritzoe D, Kaelen M, Ferguson B, De Meer I, Tanner M, Bloomfield M, Williams TM, Bolstridge M, Stewart L, Morgan CJ, Newbould RD, Feilding A, Curran HV, Nutt DJ. The effect of acutely administered MDMA on subjective and BOLD-fMRI responses to favourite and worst autobiographical memories. Int J Neuropsychopharmacol. 2014 Apr;17(4):527-40. doi: 10.1017/S1461145713001405. Epub 2013 Dec 17. PMID 24345398
- [Background] Hysek CM, Domes G, Liechti ME. MDMA enhances "mind reading" of positive emotions and impairs "mind reading" of negative emotions. Psychopharmacology (Berl). 2012 Jul;222(2):293-302. doi: 10.1007/s00213-012-2645-9. Epub 2012 Jan 27. PMID 22277989
- [Background] Kirkpatrick MG, Lee R, Wardle MC, Jacob S, de Wit H. Effects of MDMA and Intranasal oxytocin on social and emotional processing. Neuropsychopharmacology. 2014 Jun;39(7):1654-63. doi: 10.1038/npp.2014.12. Epub 2014 Jan 22. PMID 24448644
- [Background] Hysek CM, Schmid Y, Simmler LD, Domes G, Heinrichs M, Eisenegger C, Preller KH, Quednow BB, Liechti ME. MDMA enhances emotional empathy and prosocial behavior. Soc Cogn Affect Neurosci. 2014 Nov;9(11):1645-52. doi: 10.1093/scan/nst161. Epub 2013 Oct 4. PMID 24097374
- [Background] Wardle MC, de Wit H. MDMA alters emotional processing and facilitates positive social interaction. Psychopharmacology (Berl). 2014 Oct;231(21):4219-29. doi: 10.1007/s00213-014-3570-x. Epub 2014 Apr 12. PMID 24728603
- [Background] Baggott MJ, Kirkpatrick MG, Bedi G, de Wit H. Intimate insight: MDMA changes how people talk about significant others. J Psychopharmacol. 2015 Jun;29(6):669-77. doi: 10.1177/0269881115581962. Epub 2015 Apr 28. PMID 25922420
- [Background] Baggott MJ, Coyle JR, Siegrist JD, Garrison KJ, Galloway GP, Mendelson JE. Effects of 3,4-methylenedioxymethamphetamine on socioemotional feelings, authenticity, and autobiographical disclosure in healthy volunteers in a controlled setting. J Psychopharmacol. 2016 Apr;30(4):378-87. doi: 10.1177/0269881115626348. Epub 2016 Feb 15. PMID 26880224
- [Background] Carhart-Harris RL, Murphy K, Leech R, Erritzoe D, Wall MB, Ferguson B, Williams LT, Roseman L, Brugger S, De Meer I, Tanner M, Tyacke R, Wolff K, Sethi A, Bloomfield MA, Williams TM, Bolstridge M, Stewart L, Morgan C, Newbould RD, Feilding A, Curran HV, Nutt DJ. The Effects of Acutely Administered 3,4-Methylenedioxymethamphetamine on Spontaneous Brain Function in Healthy Volunteers Measured with Arterial Spin Labeling and Blood Oxygen Level-Dependent Resting State Functional Connectivity. Biol Psychiatry. 2015 Oct 15;78(8):554-62. doi: 10.1016/j.biopsych.2013.12.015. Epub 2014 Jan 10. PMID 24495461
- [Background] Liechti ME, Vollenweider FX. Which neuroreceptors mediate the subjective effects of MDMA in humans? A summary of mechanistic studies. Hum Psychopharmacol. 2001 Dec;16(8):589-598. doi: 10.1002/hup.348. PMID 12404538
- [Background] Ramos L, Hicks C, Kevin R, Caminer A, Narlawar R, Kassiou M, McGregor IS. Acute prosocial effects of oxytocin and vasopressin when given alone or in combination with 3,4-methylenedioxymethamphetamine in rats: involvement of the V1A receptor. Neuropsychopharmacology. 2013 Oct;38(11):2249-59. doi: 10.1038/npp.2013.125. Epub 2013 May 16. PMID 23676791
- [Background] Heinrichs M, Domes G. Neuropeptides and social behaviour: effects of oxytocin and vasopressin in humans. Prog Brain Res. 2008;170:337-50. doi: 10.1016/S0079-6123(08)00428-7. PMID 18655894
- [Background] Dumont GJ, Sweep FC, van der Steen R, Hermsen R, Donders AR, Touw DJ, van Gerven JM, Buitelaar JK, Verkes RJ. Increased oxytocin concentrations and prosocial feelings in humans after ecstasy (3,4-methylenedioxymethamphetamine) administration. Soc Neurosci. 2009;4(4):359-66. doi: 10.1080/17470910802649470. PMID 19562632
- [Background] Thompson MR, Hunt GE, McGregor IS. Neural correlates of MDMA ("Ecstasy")-induced social interaction in rats. Soc Neurosci. 2009;4(1):60-72. doi: 10.1080/17470910802045042. Epub 2008 May 23. PMID 18633827
- [Background] Kirkpatrick MG, Francis SM, Lee R, de Wit H, Jacob S. Plasma oxytocin concentrations following MDMA or intranasal oxytocin in humans. Psychoneuroendocrinology. 2014 Aug;46:23-31. doi: 10.1016/j.psyneuen.2014.04.006. Epub 2014 Apr 19. PMID 24882155
- [Background] Kamilar-Britt P, Bedi G. The prosocial effects of 3,4-methylenedioxymethamphetamine (MDMA): Controlled studies in humans and laboratory animals. Neurosci Biobehav Rev. 2015 Oct;57:433-46. doi: 10.1016/j.neubiorev.2015.08.016. Epub 2015 Sep 25. PMID 26408071
- [Background] Parrott AC. The psychotherapeutic potential of MDMA (3,4-methylenedioxymethamphetamine): an evidence-based review. Psychopharmacology (Berl). 2007 Apr;191(2):181-93. doi: 10.1007/s00213-007-0703-5. Epub 2007 Feb 13. PMID 17297639
- [Background] Quirk GJ, Mueller D. Neural mechanisms of extinction learning and retrieval. Neuropsychopharmacology. 2008 Jan;33(1):56-72. doi: 10.1038/sj.npp.1301555. Epub 2007 Sep 19. PMID 17882236
- [Background] Mueller D, Porter JT, Quirk GJ. Noradrenergic signaling in infralimbic cortex increases cell excitability and strengthens memory for fear extinction. J Neurosci. 2008 Jan 9;28(2):369-75. doi: 10.1523/JNEUROSCI.3248-07.2008. PMID 18184779
- [Background] Southwick SM, Bremner JD, Rasmusson A, Morgan CA 3rd, Arnsten A, Charney DS. Role of norepinephrine in the pathophysiology and treatment of posttraumatic stress disorder. Biol Psychiatry. 1999 Nov 1;46(9):1192-204. doi: 10.1016/s0006-3223(99)00219-x. PMID 10560025
- [Background] Bailey CR, Cordell E, Sobin SM, Neumeister A. Recent progress in understanding the pathophysiology of post-traumatic stress disorder: implications for targeted pharmacological treatment. CNS Drugs. 2013 Mar;27(3):221-32. doi: 10.1007/s40263-013-0051-4. PMID 23483368
- [Background] Connor TJ. Methylenedioxymethamphetamine (MDMA, 'Ecstasy'): a stressor on the immune system. Immunology. 2004 Apr;111(4):357-67. doi: 10.1111/j.0019-2805.2004.01847.x. PMID 15056370
- [Background] Ekman, P. and W.V. Friesen, Measuring facial movement. Environmental psychology and nonverbal behavior, 1976. 1(1): p. 56-75.
- [Background] Harris RJ, Young AW, Andrews TJ. Morphing between expressions dissociates continuous from categorical representations of facial expression in the human brain. Proc Natl Acad Sci U S A. 2012 Dec 18;109(51):21164-9. doi: 10.1073/pnas.1212207110. Epub 2012 Dec 3. PMID 23213218
- [Background] Dziobek I, Rogers K, Fleck S, Bahnemann M, Heekeren HR, Wolf OT, Convit A. Dissociation of cognitive and emotional empathy in adults with Asperger syndrome using the Multifaceted Empathy Test (MET). J Autism Dev Disord. 2008 Mar;38(3):464-73. doi: 10.1007/s10803-007-0486-x. Epub 2007 Nov 8. PMID 17990089
- [Background] Cami J, Farre M, Mas M, Roset PN, Poudevida S, Mas A, San L, de la Torre R. Human pharmacology of 3,4-methylenedioxymethamphetamine ("ecstasy"): psychomotor performance and subjective effects. J Clin Psychopharmacol. 2000 Aug;20(4):455-66. doi: 10.1097/00004714-200008000-00010. PMID 10917407
- [Background] Dumont GJ, Verkes RJ. A review of acute effects of 3,4-methylenedioxymethamphetamine in healthy volunteers. J Psychopharmacol. 2006 Mar;20(2):176-87. doi: 10.1177/0269881106063271. PMID 16510476
- [Background] Vollenweider FX, Gamma A, Liechti M, Huber T. Psychological and cardiovascular effects and short-term sequelae of MDMA ("ecstasy") in MDMA-naive healthy volunteers. Neuropsychopharmacology. 1998 Oct;19(4):241-51. doi: 10.1016/S0893-133X(98)00013-X. PMID 9718588
- [Background] Liechti ME, Gamma A, Vollenweider FX. Gender differences in the subjective effects of MDMA. Psychopharmacology (Berl). 2001 Mar 1;154(2):161-8. doi: 10.1007/s002130000648. PMID 11314678
- [Background] Kuypers KP, Ramaekers JG. Transient memory impairment after acute dose of 75mg 3.4-Methylene-dioxymethamphetamine. J Psychopharmacol. 2005 Nov;19(6):633-9. doi: 10.1177/0269881105056670. PMID 16272186
- [Background] Grob CS, Danforth AL, Chopra GS, Hagerty M, McKay CR, Halberstadt AL, Greer GR. Pilot study of psilocybin treatment for anxiety in patients with advanced-stage cancer. Arch Gen Psychiatry. 2011 Jan;68(1):71-8. doi: 10.1001/archgenpsychiatry.2010.116. Epub 2010 Sep 6. PMID 20819978